CLINICAL TRIAL: NCT06481280
Title: Cow's Milk Allergy (CMA): Evaluation of Tolerance, Efficacy and Safety of a Thickened Extensively Hydrolyzed Formula in Infants With IgE and Non-IgE Mediated CMA
Brief Title: Evaluation of Tolerance, Efficacy and Safety of an Hydrolyzed Formula in Infants With IgE/Non-IgE Mediated CMA.
Acronym: MERLIN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: United Pharmaceuticals (Industry)
Collaborators: Slb Pharma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: UP2022-01-MERLIN
Record Dates: First submitted 2024-06-20; First posted 2024-07-01 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Cow's Milk Allergy
Keywords: CMA (Cow's Milk Allergy); DBPCFC (Double-Blind Placebo-Controlled Food Challenge); FA (Food Allergy); IgE (Immunoglobulin E); OFC (Oral Food Challenge)
MeSH Terms: conditions — Milk Hypersensitivity; Food Hypersensitivity; Epilepsy, Idiopathic Generalized; Orofacial Cleft 1

STUDY DESIGN:
Intervention Model Description: The first part of the study consists in a double-blind placebo-controlled food challenge (DBPCFC) during which all patient will receive the test formula and a placebo, in a randomised order.
  During the second part of the study, all patients will be fed the test formula (open-label phase).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Masking only applies to the 1st part of the study : during this part all parties (participant, care provide, investigator and outcomes assessor) will be blinded.
  The 2nd study part is open-label , there is no masking during this phase
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Formula (Experimental): Infants will receive an extensively hydrolyzed formula during the double-blind placebo-controlled food challenge (DBPCFC) and will continue on this formula during the open-label feeding phase if they tolerate it.
  Interventions: Dietary Supplement: Test Formula; Dietary Supplement: Placebo Formula
- Placebo Formula (Placebo Comparator): Infants will receive a placebo formula (=their previous formula) during the DBPCFC to compare against the test formula.
  Interventions: Dietary Supplement: Test Formula; Dietary Supplement: Placebo Formula

INTERVENTIONS:
Dietary Supplement: Test Formula — Infants will receive an extensively hydrolyzed formula during the double-blind placebo-controlled food challenge (DBPCFC) and will continue on this formula during the open-label feeding phase if they tolerate it.
Dietary Supplement: Placebo Formula — Infants will receive a placebo formula during the DBPCFC to compare against the test formula.

SUMMARY:
The aim of this interventional study is to assess the hypoallergenicity of a new formula in infants having a cow milk allergy (CMA), whatever the type of CMA, meaning in both IgE-mediated and non-IgE-mediated CMA patients.

This will be tested through a double-blind placebo controlled food challenge (DBPCFC) taking place over 2 or 3 separate days, in hospital.

If the child tolerates the tested formula during the DBPCFC, he will be fed with the test formula during the second study phase. There will be monthly visit and parents will be asked to fill in diaries.

DETAILED DESCRIPTION:
Briefly, on two separate days, the placebo formula and the TEHCF will be introduced at increasing doses under medical supervision, and appearance of allergic symptoms will be witnessed and recorded if any. The week after, and more particularly the 72 hours after each food challenge day, child's parents will be instructed to report to the investigator any delayed reaction that may occur. In case the TEHCF induces an allergic reaction, the child's participation will be ended. Otherwise, the child will enter the second study part, lasting 4 months and during which the usual formula taken by the child will be totally replaced by the TEHCF.

ELIGIBILITY:
Inclusion Criteria:

* between 1 and 24 months old
* having a CMA proven in the last 3 months prior to inclusion
* free of clinical allergic symptoms for at least one week (i.e., successfully fed an elimination diet)
* whose parent(s)/legal guardian(s) signed the informed consent form.

Main Exclusion Criteria:

* Children mainly (>1 breastfeeding/day) or exclusively breastfed, with maternal willingness to continue breast-feeding
* Children with a mean formula intake lower than 250 ml/day
* Children with past anaphylactic reaction(s)
* Children with chronic (non acute) FPIES

  -- Children presenting with any situation which, according to the investigator, may interfere with the study participation, or lead to a particular risk for the subject,
* Children already participating in another clinical trial

Ages: 1 Month to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2024-08-14 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Hypoallergenicity of the formula | 7 days
  the percentage of children tolerating the formula during the double blind placebo controlled food challenge

SECONDARY OUTCOMES:
Cow's Milk Related Symptom Score (CoMiSS™) | At each visit : day7, day 30, day 60, day 90 and day 120
  The Cow's Milk Related Symptom Score (CoMiSS™) will be evaluated globally and each of its subscore. CoMiSS ranges from 0 to 33 (worst outcome).
Atopic dermatitis severity - SCORing Atopic Dermatitis (SCORAD) Index | At each visit : day7, day 30, day 60, day 90 and day 120
  Atopic dermatitis is assessed using the SCORing Atopic Dermatitis (SCORAD) Index. The score ranges from 0 to 103 (most severe state) and is used to determine the stages of severity of AD.
Gastrointestinal CMA symptoms | At each visit : day7, day 30, day 60, day 90 and day 120
  the other Gastrointestinal CMA symptoms (not described by the COMISS) will be reported (such as acute diarrhea, constipation...)
Cutaneous CMA symptoms | At each visit : day7, day 30, day 60, day 90 and day 120
  Others Cutaneous CMA symptoms besides those evaluated in the CoMISS and the SCORAD will be described
Sleep characteristics | At each visit : day7, day 30, day 60, day 90 and day 120
  This measures focuses on evaluating the quality and duration of sleep in children consuming the test.
Weight | At each monthly visit day 30, day 60, day 90 and day 120
  Weight will be expressed in kg and in z scores according to the World Health Organization (WHO) Child Growth Standards.
Height | At each monthly visit day 30, day 60, day 90 and day 120
  Height will be expressed in cm and in z scores according to the WHO Child Growth Standards.
Head circumference | At each monthly visit day 30, day 60, day 90 and day 120
  Head circumference will be expressed in cm and in z scores according to the WHO Child Growth Standards.
BMI | At each monthly visit day 30, day 60, day 90 and day 120
  BMI will be expressed in value and z scores according to the WHO Child Growth Standards.
Adverse event | During the whole study duration
  Any untoward medical reaction occuring from the signatture of the consent until the end of the participant's participation
Compliance | At each visit : day7, day 30, day 60, day 90 and day 120
  It will be assessed through the volume of formula consumed
Parents' satisfaction | At each visit : day7, day 30, day 60, day 90 and day 120
  Satisfaction regarding the effect of the study formula on regurgitations, stool consistency, digestive comfort, and the acceptability of the formula by the child will be evaluated by using a 5-level satisfaction scale (very satisfied/satisfied/unsatisfied/very unsatisfied / without opinion)
Investigator's satisfaction | At each visit : day7, day 30, day 60, day 90 and day 120
  paediatrician's satisfaction with the effect of the study formula on the child) will be assessed by using a 4-level satisfaction scale (very satisfied/satisfied/unsatisfied/very unsatisfied).
Digestive tolerance | At each visit : day7, day 30, day 60, day 90 and day 120
  Digestive tolerance of the formula will be assessed by monitoring stool frequency and consistency, regurgitations, abdominal pain/painful flatus/ bloating, crying time, irritability time.

CONTACTS AND LOCATIONS:
Overall Officials: Salvatore OLIVA, MD, PhD, Principal Investigator — University Hospital - Umberto I
Locations (2):
- Private practice Elena BRADATAN, Namur, Begium, Belgium
- University Hospital - Umberto I Sapienza, Roma, Italy

IPD SHARING:
Plan to Share IPD: No